CLINICAL TRIAL: NCT02494440
Title: Automated Fetal Femur Length Measurement by Five-Dimensional Ultrasound
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rehab Mohamed Abdelrahman, Rehab Mohamed Abdelrahman, Ain Shams University
Other Study IDs: 5D LB
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Results first posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: Automated Fetal Femur Length Measurement by Five-Dimensional Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study to evaluate Five-Dimensional Ultrasound in automated measurement of the fetal femur length at third trimester of pregnancy.

DETAILED DESCRIPTION:
This is a Prospective pilot study that will be performed at the Fetal Care Unit at Ain Shams University Maternity Hospital.

Ninety pregnant women will be recruited from the the Fetal Care Unit who will fulfill the inclusion criteria. They will be counseled to be included into the study.

All cases will be subjected to:

1. Full history taking including patient's age, parity, last menstrual period, estimated gestational age by dates, past history of medical disorders, clinical examinations (General and abdominal).
2. Two-Dimensional Ultrasound and Five-Dimensional Ultrasound will be done for all cases for assessment of fetal femur length .

The FL at Two-Dimensional Ultrasound (Gold standard) will be made from the center of the 'U' shape at each end of the bone.

The FL at Five-Dimensional Ultrasound will be measured by Pressing Five-Dimensional Ultrasound long bone Button to extract Fetal Long Bones automatically.

The estimation of gestational age by femur length by Two-Dimensional Ultrasound and Five-Dimensional Ultrasound will be compared to gestational age calculated by accurate dates of the last menstrual period.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy.
2. At third trimester of pregnancy.
3. The patient must be sure of her last normal menstrual period, last three regular cycles and no hormonal contraception before pregnancy.

Exclusion Criteria:

1. Multiple pregnancies.
2. Fetal anomalies.
3. Amniotic fluid index < 5 cm.
4. Medical disorder as diabetes mellitus, hypertension.
5. Obese patients. BMI > 30
6. Intrauterine growth retardation.
7. Post term pregnancy > 41 weeks.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This is a Prospective pilot study that will be performed at the Fetal Care Unit at Ain Shams University Maternity Hospital.
  Ninety pregnant women will be recruited from the the Fetal Care Unit who will fulfill the inclusion criteria. They will be counseled to be included into the study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
Automated Fetal Femur Length Measurement by Five-Dimensional Ultrasound

RESULTS

PARTICIPANT FLOW:
Recruitment Details: study that was performed at the Fetal Care Unit at Ain Shams University Maternity Hospital from march 2015 to march 2016.
  Ninety pregnant women were recruited from the the Fetal Care Unit who fulfilled the inclusion criteria. They were counseled and after consenting were included into the study.
Groups:
- Pregnant Women at Third Trimester of Pregnancy: 1. Two-Dimensional Ultrasound and Five-Dimensional Ultrasound were done for all cases for assessment of fetal femur length.
  2. The estimation of gestational age by femur length by Two-Dimensional Ultrasound and Five-Dimensional Ultrasound were compared to gestational age calculated by accurate dates of the last menstrual period.
Period: Overall Study
Arm/Group | Pregnant Women at Third Trimester of Pregnancy
Started | 90
Completed | 90
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Ninety pregnant women were recruited from the the Fetal Care Unit who fulfilled the inclusion criteria
Arm/Group | Pregnant Women at Third Trimester of Pregnancy
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 90
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 0
Region of Enrollment [Number; unit: participants]
  Egypt | 90

OUTCOME MEASURES:

1. Primary Outcome: Gestational Age Calculated by Accurate Dates of the Last Menstrual Period
Description: The patient must be sure of her last normal menstrual period, last three regular cycles and no hormonal contraception before pregnancy.
  Gestational age calculated by the last menstrual period
Time Frame: 26 - 40 weeks of gestation
Population: 90 pregnant women were recruited from the the Fetal Care Unit who fulfilled the inclusion criteria
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Pregnant Women at Third Trimester of Pregnancy
Number analyzed (Participants) | 90
weeks | 35.6 (3.4)

2. Secondary Outcome: Gestational Age Calculated by Femur Length Measurement by Two-Dimensional Ultrasound
Description: The femur length at Two-Dimensional Ultrasound (Gold standard) was made from the center of the 'U' shape at each end of the bone. After the long axis of the fetus was identified, the transducer was turned 90 degrees to produce a cross sectional image of fetal trunk, maintaining the 90 degrees angle until the lower spine and iliac crest were identified, then the transducer was rotated until a full femur was imaged. The femur length was measured from the center of the "U" shape at each end of the bone; this represented the length of the metaphysis).
  then , Gestational Age Calculated by femur length measurement
Time Frame: 26 - 40 weeks of gestation
Population: 90 pregnant women were recruited from the the Fetal Care Unit who fulfilled the inclusion criteria
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Pregnant Women at Third Trimester of Pregnancy
Number analyzed (Participants) | 90
weeks | 33.4 (2.8)

3. Secondary Outcome: Gestational Age Calculated by Femur Length Measurement by Five-Dimensional Ultrasound
Description: The femur length at Five-Dimensional Ultrasound: To obtain 3D volume data, the entire bone length of the femur was identified on the screen, as in the 2D-ultrasound measurement, and the long axis of the femur was placed in the direction of the x axis in the image in which the ultrasound beam was perpendicular to the bone. The 5D LB set key was pressed on the system, wherein the system automatically analyzed the 3D volume data, reconstructed the 3D image of the long bones, and displayed the measured length of the femur length on the screen was measured by pressing 5D LB Button to extract Fetal Long Bones automatically.
  then, gestational Age Calculated by femur length measurement
Time Frame: 26 - 40 weeks of gestation
Population: Ninety pregnant women were recruited from the the Fetal Care Unit who fulfilled the inclusion criteria
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Pregnant Women at Third Trimester of Pregnancy
Number analyzed (Participants) | 90
weeks | 33.4 (2.9)

ADVERSE EVENTS:
Time Frame: 1 year from march 2015 to march 2016
Description: Two-Dimensional Ultrasound and Five-Dimensional Ultrasound were performed and adverse Events Adverse Events were assessed.
Arm/Group | Pregnant Women at Third Trimester of Pregnancy
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No